CLINICAL TRIAL: NCT04619940
Title: Validity and Reliability of iPhone Application in Active Internal Rotation Measurement of Shoulder in Patients With Shoulder Pain
Brief Title: Validity and Reliability of iPhone Application in Internal Rotation Measurement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Bilinç Doğruöz Karatekin, MD, Specialist of PMR, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: IMU Shoulder
Record Dates: First submitted 2020-10-29; First posted 2020-11-06 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Shoulder Pain
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Intervention Model Description: Measurements were conducted separately in different cabinets without seeing each other for each participant by 1 physical medicine and rehabilitation specialist and 1 physiotherapist. The measurements were recorded in separate locations until all participants were completed.
Who Masked: Investigator
Masking Description: Measurements were conducted separately in different cabinets without seeing each other for each participant by 1 physical medicine and rehabilitation specialist and 1 physiotherapist. The measurements were recorded in separate locations until all participants were completed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iHandy application (Experimental): The IHandy® app is a free app with a visual display similar to that of the digital inclinometer in terms of digital size. In this study, due to its prevalence in the literature and its use in clinics, manual goniometer (gold standard) was chosen to be compared with this iPhone application.
  Interventions: Diagnostic Test: iHandy application; Diagnostic Test: Standard Goniometer
- Standard goniometer (Active Comparator): While measuring with goniometer, the pivot point of the goniometer was placed on the olecranon, the immobile rod of the goniometer was kept parallel to the bed, while the moving rod was kept parallel to the ulna, the angle was recorded at the end point of the movement.
  Interventions: Diagnostic Test: iHandy application; Diagnostic Test: Standard Goniometer

INTERVENTIONS:
Diagnostic Test: iHandy application — The IHandy® app is a free app with a visual display similar to that of the digital inclinometer in terms of digital size. In this study, due to its prevalence in the literature and its use in clinics, manual goniometer (gold standard) was chosen to be compared with this iPhone application.
Diagnostic Test: Standard Goniometer — While measuring with goniometer, the pivot point of the goniometer was placed on the olecranon, the immobile rod of the goniometer was kept parallel to the bed, while the moving rod was kept parallel to the ulna, the angle was recorded at the end point of the movement.

SUMMARY:
The validity and reliability of active internal rotation ROM measurement of shoulder with smartphone in patients with shoulder pain was investigated.

DETAILED DESCRIPTION:
Eighteen patients with shoulder pain who applied to the Physical Medicine and Rehabilitation, shoulder subspecialty outpatient clinic who agreed to participate in the study and 18 volunteers who had not experienced shoulder pain before enrolled in the study. Participant age range was determined as 40-70 years.

The IHandy® app is a free app with a visual display similar to that of the digital inclinometer in terms of digital size. In this study, due to its prevalence in the literature and its use in clinics, manual goniometer (gold standard) was chosen to be compared with this iPhone application.

The participants were asked to lie on the bed in supine position with shoulder to be measured at the edge of the bed. The measured shoulder was positioned at 90 degrees abduction, 90 degrees elbow flexion and forearm at neutral position. The participant was asked to bring the wrist closer to the bed in the direction of the little finger, and was measured at the angle that the shoulder could not move without lifting the arm. In the measurement made with the application, the phone was held parallel to the ulna and the value displayed on the screen was recorded. The participant were asked to repeat the movement if his/her shoulder lift up of bed, straightened his/her elbow, or did anything that would disrupt her movement pattern.

Each measurement was repeated 3 times and after 2 weeks the control measurements were made by repeating 3 times.

Measurements were conducted separately in different cabinets without seeing each other for each participant by 1 physical medicine and rehabilitation specialist and 1 physiotherapist. The measurements were recorded in separate locations until all participants were completed.

ELIGIBILITY:
Inclusion Criteria:

* Patient with shoulder pain
* 40-70 years old
* Agreed to participate the study

Exclusion Criteria:

* <40 years old or >70 years old
* Not agreed to participate

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
iHandy application | 6 months
  The IHandy® app is a free app with a visual display similar to that of the digital inclinometer. In the measurement made with the application, the phone was held parallel to the ulna and the value displayed on the screen was recorded as range of motion value.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medeniyet University Faculty of Medicine, Physical Medicine and Rehabilitation Department, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided